CLINICAL TRIAL: NCT00075348
Title: Genetic Mutation Analysis In A VHL Population
Brief Title: Genetic Study to Identify Gene Mutations in Participants Previously Enrolled in Clinical Trial NCI-99-C-0053 Who Have Von Hippel-Lindau Syndrome or Are at Risk for Von Hippel-Lindau Syndrome
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: 030148; 03-C-0148; CDR0000302478
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Kidney Cancer; Von Hippel-lindau Syndrome
Keywords: renal cell carcinoma; von Hippel-Lindau syndrome
MeSH Terms: conditions — Kidney Neoplasms; von Hippel-Lindau Disease; Carcinoma, Renal Cell

INTERVENTIONS:
Genetic: mutation analysis

SUMMARY:
RATIONALE: The identification of gene mutations in individuals who have or are at risk for von Hippel-Lindau syndrome may allow doctors to better determine the genetic processes involved in the development of cancer.

PURPOSE: This genetic study is finding gene mutations in participants with von Hippel-Lindau syndrome or who are at risk for developing von Hippel-Lindau syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Obtain laboratory identification and confirmation of research results for gene mutations in participants previously enrolled in NCI-99-C-0053 who have von Hippel-Lindau (VHL) syndrome or who are at risk for VHL syndrome.
* Determine genotype status in these participants.

OUTLINE: Participants submit a blood or buccal sample for genetic mutation analysis. Participants may receive genetic counseling and/or the results of genetic testing, if desired.

PROJECTED ACCRUAL: A maximum of 260 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Prior enrollment in the von Hippel-Lindau (VHL) Syndrome Epidemiology Study NCI-99-C-0053
* Meets 1 of the following criteria:

  * Diagnosis of VHL syndrome
  * At risk of VHL syndrome
  * Family member of patient with VHL syndrome
* VHL syndrome genotype is not known

PATIENT CHARACTERISTICS:

Age

* Adult

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2003-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William M. Linehan, MD, Study Chair — NCI - Urologic Oncology Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States